CLINICAL TRIAL: NCT00127049
Title: A Prospective Multicenter Phase II Trial of Gemcitabine, Cisplatin, and Ifosfamide (GIP) in Patients With Relapsed Non-Seminomatous Germ-Cell Tumors (NSGCT) and a Predicted Favorable Prognosis
Brief Title: Trial of Gemcitabine, Cisplatin, and Ifosfamide in Patients With Relapsed Non-Seminomatous Germ-Cell Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIP-TG
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Germ Cell Tumor
Keywords: Patients with relapsed non-seminomatous germ-cell tumors (NSGCT)
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Gemcitabine; Ifosfamide; Cisplatin; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: gemcitabine, ifosfamide, cisplatin, G-CSF

SUMMARY:
This is a prospective multicenter phase II trial of gemcitabine, cisplatin, and ifosfamide (GIP) in patients with relapsed non-seminomatous germ-cell tumors (NSGCT) and a predicted favorable prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 16 years
* Histologically-proven disseminated (non stage I) NSGCT, or diagnosis of NSGCT based on very elevated serum human chorionic gonadotropin (HCG) and/or alpha fetoprotein (AFP)
* Relapsed disease classified as good prognosis according to the Memorial Sloan-Kettering Cancer Center (MSKCC) classification criteria:

  * Testicular primary site
  * Prior treatment limited to one program (or 6 or fewer cycles of cisplatin)
  * Either a complete response or a partial response with normal serum AFP and HCG
* Relapse documented by rising AFP and/or HCG or by a biopsy
* No previous carcinoma, except basal-cell carcinoma of the skin
* Adequate renal function: measured or calculated creatinine clearance> 60 ml/min
* Absolute granulocyte count >= 1,500/mm3, platelets >= 100,000 mm3, bilirubin < 1.5 fold the upper normal value
* Signed informed consent.

Exclusion Criteria:

* Patients infected by the human immunodeficiency virus (HIV)
* Patients who do not fit inclusion criteria

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37
Dates: Start 2004-12

PRIMARY OUTCOMES:
Complete response rate

SECONDARY OUTCOMES:
Toxicity
Progression free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Fizazi K, Gravis G, Flechon A, Geoffrois L, Chevreau C, Laguerre B, Delva R, Eymard JC, Rolland F, Houede N, Laplanche A, Burcoveanu D, Culine S. Combining gemcitabine, cisplatin, and ifosfamide (GIP) is active in patients with relapsed metastatic germ-cell tumors (GCT): a prospective multicenter GETUG phase II trial. Ann Oncol. 2014 May;25(5):987-91. doi: 10.1093/annonc/mdu099. Epub 2014 Mar 4. PMID 24595454